CLINICAL TRIAL: NCT03043404
Title: REPRISE II FLEX: Repositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of LotuS™ ValvE With a FLEXible Delivery System - Confirmation of Performance and Safety
Brief Title: Performance and Safety of the Lotus™ Valve With a FLEXible Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2321
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lotus Valve Flex System (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve FLEX System
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — TAVR with Lotus Valve Flex System

SUMMARY:
To confirm the acute performance and safety of the Lotus™ Valve Flex System for transcatheter aortic valve replacement (TAVR) in symptomatic patients with severe calcific aortic stenosis who are considered high risk for surgical valve replacement.

DETAILED DESCRIPTION:
This clinical study is a prospective, single-arm study designed to confirm that the acute performance and safety of the Lotus Valve Flex System for TAVR are consistent with the results of the Lotus Valve System in the REPRISE II study, when delivered and deployed in symptomatic subjects who have severe calcific aortic valve stenosis and who are at high risk for surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is ≥70 years of age
* 2. Subject has documented calcific native aortic valve stenosis with an initial aortic valve area (AVA) of <1.0 cm2 (or AVA index of <0.6 cm2/m2) and either a mean pressure gradient >40 mm Hg or a jet velocity >4 m/s, as measured by echocardiography
* 3. Subject has a documented aortic annulus size between ≥20 and ≤27 mm based on pre-procedure diagnostic imaging
* 4. Symptomatic aortic valve stenosis with NYHA Functional Class ≥ II
* 5. Subject is considered high risk for surgical valve replacement based on at least one of the following:

  1. Society of Thoracic Surgeons (STS) score ≥8%, AND/OR
  2. Agreement by the heart team (which must include an in-person evaluation by an experienced cardiac surgeon) that subject is at high operative risk of serious morbidity or mortality with surgical valve replacement
* 6. Heart team (which must include an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement.
* 7. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
* 8. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

1. Subject has a congenital unicuspid or bicuspid aortic valve.
2. Subject with an acute myocardial infarction within 30 days of the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).
3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months, or has any permanent neurologic defect prior to study enrollment.
4. Subject is on dialysis or has serum creatinine level >3.0 mg/dL or 265 µmol/L.
5. Subject has a pre-existing prosthetic heart valve (aortic or mitral) or a prosthetic ring in any position.
6. Subject has ≥3+ mitral regurgitation, ≥3+ aortic regurgitation or ≥3+ tricuspid regurgitation (i.e., subject cannot have more than moderate mitral, aortic or tricuspid regurgitation).
7. Subject has a need for emergency surgery for any reason.
8. Subject has a history of endocarditis within 12 months of index procedure or evidence of an active systemic infection or sepsis.
9. Subject has echocardiographic evidence of intra-cardiac mass, thrombus or vegetation.
10. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
11. Subject requires chronic anticoagulation therapy (warfarin) and cannot tolerate concomitant therapy with either aspirin or clopidogrel.

    Note: Subjects who require chronic anticoagulation must be able to be treated additionally with either aspirin or clopidogrel. An alternative P2Y12 inhibitor may be prescribed if subject is allergic to or intolerant of clopidogrel.
12. Subject has active peptic ulcer disease or gastrointestinal bleed within the past 3 months, other bleeding diathesis or coagulopathy or will refuse transfusions.
13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all thienopyridines, heparin, nickel, tantalum, titanium, or polyurethanes.
14. Subject has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrollment.
15. Subject has hypertrophic obstructive cardiomyopathy.
16. Subject has any therapeutic invasive cardiac procedure (including balloon aortic valvuloplasty) within 30 days prior to the index procedure (except for pacemaker implantation which is allowed).
17. Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization.
18. Subject has documented left ventricular ejection fraction <30%.
19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
20. Subject has severe peripheral vascular disease (including aneurysm defined as maximal luminal diameter >5 cm or with documented presence of thrombus, marked tortuosity, narrowing of the abdominal aorta, severe unfolding of the thoracic aorta or thick [>5 mm], protruding or ulcerated atheroma in the aortic arch) or symptomatic carotid or vertebral disease.
21. Femoral artery lumen of <6.0 mm for subjects requiring 23 mm valve size or <6.5 mm for subjects requiring 27 mm valve size, or severe iliofemoral tortuosity or calcification that would prevent safe placement of the introducer sheath.
22. Current problems with substance abuse (e.g., alcohol, etc.).
23. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
24. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Technical success | immediately post-procedure
  defined as successful vascular access, delivery and deployment of the Lotus Valve and successful retrieval of the delivery system; and correct positioning of a single Lotus Valve in the proper anatomical location; reported as percent of subjects.

SECONDARY OUTCOMES:
Mean aortic valve pressure gradient and effective orifice area | at discharge or 7 days post-procedure (whichever comes first)
  as measured by echocardiography and assessed by an independent core laboratory
Device performance | at discharge or 7 days post-procedure (whichever comes first)
  defined as successful repositioning of the Lotus Valve if repositioning is attempted; and successful retrieval of the Lotus Valve if retrieval is attempted; and grade of paravalvular aortic regurgitation, as measured by echocardiography and assessed by an independent core laboratory

OTHER OUTCOMES:
Mortality: all-cause, cardiovascular, and non-cardiovascular | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Stroke: disabling and non-disabling | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Composite of all-cause mortality and disabling stroke | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Bleeding: life-threatening (or disabling) and major | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Myocardial infarction (MI) | periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure)
Acute kidney injury: based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2 | ≤7 days post index procedure
Major vascular complication | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV) | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
New permanent pacemaker implantation resulting from new or worsened conduction disturbances (including new left bundle branch block [LBBB] and third degree atrioventricular block) | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
New onset of atrial fibrillation or atrial flutter | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Coronary obstruction | ≤7 days post procedure
Ventricular septal perforation, reported as percent of subjects | ≤7 days post procedure
Mitral apparatus damage, reported as percent of subjects | ≤7 days post procedure
Cardiac tamponade, reported as percent of subjects | ≤7 days post procedure
Prosthetic aortic valve malposition, including valve migration, valve embolization, ectopic valve deployment, or transcatheter aortic valve (TAV)-in-TAV deployment | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Prosthetic aortic valve thrombosis | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Prosthetic aortic valve endocarditis | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Prosthetic aortic valve performance | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
  as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Functional status | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
  as evaluated by the New York Heart Association (NYHA) classification
Neurological status | at discharge and 1 year
  as determined by the National Institutes of Health Stroke Scale (NIHSS)
Neurological status | at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
  as determined by the Modified Rankin Scale (mRS)

CONTACTS AND LOCATIONS:
Overall Officials: Ian T Meredith, MD, PhD, Principal Investigator — Monash
Locations (2):
- Australia (2):
  - Prince Charles Hospital, Chermside, Queensland
  - Monash Heart, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No